CLINICAL TRIAL: NCT05619367
Title: A Compassionate Use (CU) Program of Odronextamab
Status: Available | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R1979-Odronextamab
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Relapsed or Refractory (R/R) Follicular Lymphoma (FL); Diffuse Large B-Cell Lymphoma (DLBCL); B-Cell Non-Hodgkin Lymphoma (NHL); High-Grade B-Cell Lymphoma (HGBCL)
MeSH Terms: conditions — Recurrence; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Odronextamab
  Other Names: REGN1979

SUMMARY:
Provide compassionate use of odronextamab

Sex: All
Age Groups: Child, Adult, Older Adult